CLINICAL TRIAL: NCT06188767
Title: Long-term Effects of Anabolic Androgenic Steroids on Muscle Growth Potential: Testosterone-induced Muscle Memory and Underlying Mechanisms
Brief Title: Testosterone-induced Muscle Memory and Underlying Mechanisms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Morten Hostrup, PhD (Other)
Responsible Party: Sponsor-Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TESTO
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Skeletal Muscle Physiology
MeSH Terms: interventions — testosterone undecanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone (Experimental): Participants are randomized to a single injection of 1000 mg testosterone undecanoate
  Interventions: Drug: Testosterone Undecanoate
- Placebo (Placebo Comparator): Participants are randomized to a single placebo injection
  Interventions: Drug: Testosterone Undecanoate

INTERVENTIONS:
Drug: Testosterone Undecanoate — Following testosterone/placebo injection, participants undergo supervised resistance training for 4 weeks. This period is followed by a washout period with no drug and either continued resistance training or detraining for 16 weeks. Thereafter, another 4-week period with supervised resistance training is commenced, with no drug.

SUMMARY:
The purpose of this project is to investigate underlying mechanisms of testosterone- and resistance training-induced muscle hypertrophy and muscle memory in humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* BMI of <26 and normal ECG and blood pressure

Exclusion Criteria:

* Smoking
* Chronic disease,
* Use of prescription medication
* Pain due to current or previous musculoskeletal injury
* Resistance training more than once per week in the 12 months leading up to the intervention
* Current or previous use of prohibited anabolic substances

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Fiber cross-sectional area | The change in fiber cross-sectional is assessed at baseline, 4, 20 and 24 weeks
  Immunohistochemistry to determine fiber cross-sectional area
Myonuclei | The change in myonuclei is assessed at baseline, 4, 20 and 24 weeks
  Immunohistochemistry to determine number of myonuclei
Skeletal muscle proteome | The change in the muscle proteome is assessed at baseline, 4, 20 and 24 weeks
  Pathway enrichment analysis of the muscle proteome using mass spectrometry-based proteomics

SECONDARY OUTCOMES:
Lean mass | The change in lean mass is assessed at baseline, 4, 20 and 24 weeks
  Lean mass assessed by dual X-ray absorptiometry (DXA)
Satellite cells | The change in satellite cells is assessed at baseline, 4, 20 and 24 weeks
  Immunohistochemistry to determine number of satellite cells
Muscle strength | The change in 1-repetition maximum is assessed at baseline, 4, 20 and 24 weeks
  1-repetition maximum

CONTACTS AND LOCATIONS:
Locations (1):
- The August Krogh Section for Human and Molecular Physiology, Department of Nutrition, Exercise and Sports, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided